CLINICAL TRIAL: NCT03284320
Title: Retrospective Study to Evaluate Efficacy and Safety of Trabectedin (Yondelis®) in Sarcoma Patients
Brief Title: Retrospective Study in Sarcoma Patients
Acronym: ReTraSarc
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Other Study IDs: GISG-14
Record Dates: First submitted 2017-08-21; First posted 2017-09-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Sarcoma of Bone; Sarcoma of Soft Tissue
Keywords: Drug therapy; Treatment outcome; Adult
MeSH Terms: conditions — Osteosarcoma; Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objectives of this trial is to evaluate efficacy and safety of treatment with Trabectedin in a large cohort of German patients with soft tissue and bone sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed soft tissue or bone sarcomas treated with at least one cycle of Trabectedin in any line of therapy.
* Age ≥18years at start of therapy with Trabectedin
* Informed Consent
* Patients already deceased may be included when the treating physician is able to determine the presumptive consent

Exclusion Criteria:

* No follow-up data available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with soft tissue and bone sarcomas treated with Trabectedin
Sampling Method: Non-Probability Sample
Enrollment: 514 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
- Progression free survival (PFS) | At the time of every treatment documentation up to the end of treatment, approximately 2 years
- Overall survival (OS) | At the time of every treatment documentation up to the end of treatment, approximately 2 years

SECONDARY OUTCOMES:
CTCAE (Common Terminology Criteria for Adverse Events) 4.03 | At the time of every treatment documentation up to the end of treatment, approximately 2 years
  Safety Evaluation according to toxitiy

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pink, MD, Principal Investigator — University Medicine Greifswald; Peter Reichardt, MD, Principal Investigator — Sarcoma Center Berlin-Brandenburg; HELIOS Hospital Berlin Buch
Locations (1):
- University Medicine Greifswald, Department of Internal Medicine C, Greifswald, Germany

REFERENCES:
- [Background] Pink D, Bertz-Lepel J, Busemann C, Bitz U, Reichardt P. Efficacy of trabectedin in patients with advanced or metastatic alveolar soft-part sarcoma. Onkologie. 2012;35(5):249-52. doi: 10.1159/000338342. Epub 2012 Apr 23. PMID 22868503